CLINICAL TRIAL: NCT01110941
Title: A Multicenter Feasibility Study With S-1, Oxaliplatin and Oral Leucovorin (SOL) for the Patients With Untreated Metastatic Colorectal Cancer
Brief Title: Feasibility Study of SOL (S-1,Oral Leucovorin,and Oxaliplatin) for Colorectal Cancer in China
Acronym: SCI-101
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shen Lin (Other)
Collaborators: 307 Hospital of PLA (Other); Beijing Union Hosptial (Unknown); Tianjin Medical University Cancer Institute and Hospital (Other); Hebei Provincial Cancer Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Shen Lin, pro, Peking University
Organization: Peking University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOL feasibility study
Record Dates: First submitted 2010-04-21; First posted 2010-04-27 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Colorectal Cancer
Keywords: S-1; leucovorin; oxaliplatin; colorectal cancer; SOL; unresectable or recurrent colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — S 1 (combination); Leucovorin; Oxaliplatin; Long-Term Synaptic Depression

ARMS (1):
- SOL (Experimental): single arm
  Interventions: Drug: S-1, leucovorin, oxaliplatin

INTERVENTIONS:
Drug: S-1, leucovorin, oxaliplatin — S-1(20mg、25mg), capsule, 40~60mg, Bid,p.o., day1~7； LV (25 mg), tablet, 25mg,Bid,p.o., day1~7； L-OHP (50 mg),injection 85mg/m2, day1. repeated at every 2 weeks cycle till disease progression.
  Other Names: S-1(20mg、25mg)--Taiho Pharmaceutical Co., Ltd.；; LV (25 mg)；; L-OHP (50 mg)--Sanofi Aventis Co., Ltd.

SUMMARY:
S-1 is an oral fluoropyrimidine with demonstrated efficacy on gastric cancer and colorectal cancer. The new regimen with Oxaliplatin and leucovorin is expected to achieve more encouraging efficacy on colorectal cancer. This study is to explore the feasibility of the SOL regimen on efficacy and tolerability on Chinese colorectal cancer patients.

DETAILED DESCRIPTION:
* Endpoints:
* Primary endpoints: adverse drug reaction
* Secondary endpoints:

  * Overall Response Rate：ORR
  * Progress Free Survival: PFS
  * Time to Treatment Failure：TTF

ELIGIBILITY:
Inclusion Criteria:

* Advanced unresectable or recurrent colorectal cancer patients which meet the following criteria:

  * Willing to sign ICF
  * Could orally take investigational product
  * Pathology diagnosis is adenocarcinoma
  * Above 20 years
  * No previous treatment(including: radiotherapy,chemotherapy and immunotherapy)
  * For recurrent cases, if the patient had received adjuvant chemotherapy that didn't include S-1 and L-OHP in 180 days ago, he/she could be enrolled in
  * With target lesions with diameter which is longer than 1cm in spiral CT or MRI examination within 30 days
* Lab test within 15 days meet following criteria

  * Hemoglobin higher than 9.0g/dL
  * Leukocyte higher than 12,000/mm3
  * Neutrophil higher than 2,000/mm3
  * PLT higher than 10.0 104/mm3
  * Bilirubin lower than 1.5 times of upper limit of normal range
  * AST,ALT,ALP lower than 2.5 times of upper limit of normal range
  * Creatinine lower than upper limit of normal range

When patient has liver metastasis or bone metastasis, the value of AST,ALT,ALP could be within 5 times of upper limit of normal range

* ECOG 0 or 1
* Expected survival time more than 90 days

Exclusion Criteria:

* The patient who meet the following criteria should be excluded from this trial
* Patients who have severe drug allergic history(including: platinum related drugs,5-FU,FT,LV,5-HT3 receptor antagonist)
* Attended other clinical trial within 4 weeks
* Received transfusion of blood,related products or G-CSF within 15 days
* Received surgery within 4 weeks and the effect hadn't vanished
* Have diarrhea
* Have complication of active infection(infection caused fever higher than 38℃)
* Have complication of poor controlled hypercalcemia,hypertension,diabetes
* Have complication of severe ECG abnormal or other heart disease which will affect clinical treatment(including: cardiac dysfunction,myocardial infarction,angina)
* Have complication of severe pulmonary disease(including:interstitial pneumonia,pulmonary fibrosis,severe emphysema)
* Have complication of psychiatric disorder which will affect clinical treatment or have history of CNS disease
* Have complication of active gastrointestinal bleeding
* Have pleural effusion,ascites or pericardial effusion that need drainage
* Have complication of multiple bone metastasis
* Have severe complication(including:ileus,renal insufficiency,hepatic insufficiency,cerebrovascular disturbance)
* Have brain metastasis or suspicious brain metastasis
* Have active multiple primary cancer
* Female patients who are in pregnancy or lactation and patients who are not willing to take contraception measures
* Investigator judge not eligible to this trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | from first administration till 28 days after last dosage

SECONDARY OUTCOMES:
Tumor response according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria, and follow up till disease progression or withdrawal from study due to intolerable adverse events (AE) | every 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lu M, Wang Y, Liu W, Bai C, Xu J, Shen L. A Multicenter Feasibility Study with S-1, Oxaliplatin and Oral Leucovorin (SOL) for the Patients with Untreated Metastatic Colorectal Cancer: The Result of Final Analysis. Hepatogastroenterology. 2014 Jun;61(132):1018-23. PMID 26158159